CLINICAL TRIAL: NCT02846129
Title: Incidence of Complications Associated With Anesthesia in Multiple Gestation Undergoing Cesarean Delivery: A Retrospective Review
Brief Title: Incidence of Complications Associated With Anesthesia in Multiple Gestation Undergoing Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Patchareya Nivatpumin, Assistant professor, Mahidol University
Other Study IDs: 067/2559(EC3)
Record Dates: First submitted 2016-03-13; First posted 2016-07-27 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Multiple Gestation; Cesarean Delivery; Anesthesia
Keywords: multiple gestation; complications; cesarean delivery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Incidence of anesthesia related complications in multiple gestation patients undergoing cesarean delivery has not been reported in Thailand. The aim of this study is to identify complications that occur which may derived from different anesthetic techniques used, such as hypotension, uterine atony, postpartum hemorrhage, rate of hysterectomy, blood transfusion and fetal outcome.

DETAILED DESCRIPTION:
Nowadays, the rate of multiple gestations is increasing considerably due to the prevalence of assisted reproductive technology. As physiologic changes from multiple gestations differ from singleton pregnancy, multiple gestations are considered a high risk pregnancy. A number of complications can occur from prenatal period such as preterm labor and increase rate of maternal beta agonist usage e.g. ritodrine, terbutaline and salbutamol. These drugs cause maternal tachycardia, hypokalemia and pulmonary edema. Multiple gestations increase rate of cesarean delivery and intraoperative complications such as postpartum hemorrhage and hysterectomy can be found 3.7 times and 2.3 times respectively higher than that of singleton pregnancy.

Spinal anesthesia is the anesthetic technique of choice for parturients undergoing cesarean section, owing to its rapid onset of action, reliability, superior postoperative pain control and lower mortality rate than general anesthesia. However, the most important complication is maternal hypotension, especially in multiple gestations that may derive from more aortocaval compression comparing with singleton pregnancy. Nevertheless, some patients having contraindications for regional anesthesia e.g. thrombocytopenia, coagulopathy or pulmonary edema make anesthesiologists decide to put these patients under general anesthesia for cesarean section. General anesthesia for cesarean section in singleton pregnancy has been proved that can cause higher incidence of postpartum hemorrhage and higher rate of blood transfusion compared to regional anesthesia.

Incidence of anesthesia related complications in multiple gestation patients undergoing cesarean delivery has not been reported in Thailand. The aim of this study is to identify complications that occur which may derived from different anesthetic techniques used, such as hypotension, uterine atony, postpartum hemorrhage, rate of hysterectomy, blood transfusion and fetal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, multiple gestation underwent cesarean delivery from the past until 31 Dec 2015

Exclusion Criteria:

* Preterm delivery before 24 weeks
* Death fetus in utero

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women, multiple gestation e.g. twin, triplet, quadruplet undergoing cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 1057 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of complications associated with anesthesia in multiple gestation undergoing cesarean section | Up to 24 hours postoperatively

SECONDARY OUTCOMES:
Anesthetic technique used e.g. regional or general anesthesia | Up to 24 hours postoperatively
Amount of medication used | Up to 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Bangkok, Thailand
Locations (1):
- Anesthesiology department, Siriraj hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trojner-Bregar A, Tul N, Verdenik I, Novak Z, Blickstein I. Puerperal morbidity following repeat cesarean delivery in twin pregnancies. Arch Gynecol Obstet. 2013 Sep;288(3):551-4. doi: 10.1007/s00404-013-2818-8. Epub 2013 Mar 28. PMID 23536103
- [Background] Walker MC, Murphy KE, Pan S, Yang Q, Wen SW. Adverse maternal outcomes in multifetal pregnancies. BJOG. 2004 Nov;111(11):1294-6. doi: 10.1111/j.1471-0528.2004.00345.x. PMID 15521878
- [Background] Marino T, Goudas LC, Steinbok V, Craigo SD, Yarnell RW. The anesthetic management of triplet cesarean delivery: a retrospective case series of maternal outcomes. Anesth Analg. 2001 Oct;93(4):991-5. doi: 10.1097/00000539-200110000-00039. PMID 11574371
- [Background] Rouse DJ, MacPherson C, Landon M, Varner MW, Leveno KJ, Moawad AH, Spong CY, Caritis SN, Meis PJ, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai BM, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Blood transfusion and cesarean delivery. Obstet Gynecol. 2006 Oct;108(4):891-7. doi: 10.1097/01.AOG.0000236547.35234.8c. PMID 17012451
- [Background] Butwick AJ, Carvalho B, El-Sayed YY. Risk factors for obstetric morbidity in patients with uterine atony undergoing caesarean delivery. Br J Anaesth. 2014 Oct;113(4):661-8. doi: 10.1093/bja/aeu150. Epub 2014 Jun 6. PMID 24907281